CLINICAL TRIAL: NCT02050113
Title: Complex Aortic Aneurysm Repair Using Physician Modified Endografts and Custom Made Devices
Acronym: CARPE-CMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andres Schanzer (Other)
Responsible Party: Sponsor-Investigator, Andres Schanzer, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARPE-01
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Complex Aortic Aneurysms; Thoracoabdominal Aneurysms; Pararenal Aneurysms; Juxtarenal Aneurysms; Marfan Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome; Aortic Arch Aneurysm
Keywords: Complex Aortic Aneurysms; Thoracoabdominal Aneurysms; Pararenal Aortic Aneurysms; Juxtarenal Renal Aneurysms; Endovascular Branch Graft; Fenestrated Stent Graft; Abdominal Aortic Aneurysm; Endovascular; Aortic Dissection; Aortic Arch Aneurysms
MeSH Terms: conditions — Marfan Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome; Aneurysm, Aortic Arch; Aortic Aneurysm, Abdominal; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endovascular repair (Experimental): Endovascular repair of Complex Aortic Aneurysm using a physician modified stent graft. custom made device or arch branch device.
  Interventions: Device: Custom Made Fenestrated or Branched Stent Graft

INTERVENTIONS:
Device: Custom Made Fenestrated or Branched Stent Graft — The surgeon will place a custom made graft, t-Branch device or modify commercially available stent grafts to match the anatomy of the patient being treated. Small fenestrations (holes) will be made in the stent graft so that additional stents can be inserted through the fenestration and into the blood vessels that lead to the kidneys, intestines or liver. These stents allow blood to flow freely to these organs. If the aneurysm is in the aortic arch stents may be placed in the carotid and subclavian arteries. This surgery is done through small incisions in the groin and sometimes in the upper arm.
  Other Names: t-Branch Device; Physician Modified Device; Arch Branch Device

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of custom made devices, Zenith t-Branch devices and physician modification of FDA approved off-the-shelf endovascular grafts in the treatment of patients with complex abdominal aneurysms, aortoiliac aneurysms, thoracoabdominal aneurysms and aortic arch aneurysms who (1) have anatomy not suitable for endovascular repair using grafts currently marketed in the United States,(2) are deemed unsafe to wait the required time necessary for commercial endograft manufacturing, and (3) are at high risk for open surgical repair. Amendment to the study has created a cohort open to people with connective tissue diseases such as Marfan, Ehlers-Danlos or Loey-Dietz syndromes to enroll in the trial. An additional amendment to the study allows the use of a custom made device to treat an aneurysm in the aortic arch.

DETAILED DESCRIPTION:
Endovascular repair of complex aortic aneurysms is limited by the need to maintain blood flow to the critical organs that receive blood from the aorta, such as the kidneys, liver and intestines. While there are some commercially available devices that may treat some of these patients these devices may not be suitable or available for a given patient. In this study we will use custom made devices manufactured by Cook, Inc, Zenith t-Branch devices and off-the-shelf, FDA approved devices which are altered by creating fenestrations (holes) in the stent graft that allow additional stents to be inserted into the blood vessels that supply blood to these critical organs.

Determination of which type of endograft to use will be based on the patient's anatomy and the perceived urgency of the need for repair. This decision will be made by the study team and confirmed by a 3rd party reviewer who is not an investigator on the study team. After ensuring that a patient meets inclusion and exclusion criteria for participation in the CARPE-CMD study, the perceived urgency for repair will be evaluated given the 6-8 week required time for manufacture of a CMD device.

If the patient's aneurysm is not symptomatic and if, at the discretion of the treating surgeon, the patient is deemed safe to wait 8 weeks until repair, the patient will be considered non-urgent. Non-urgent patients will undergo repair with a CMD device.

If the patient's aneurysm is symptomatic and if, at the discretion of the treating surgeon, the patient is deemed unsafe to wait 8 weeks until repair, the patient will be considered urgent. Urgent patients will undergo repair with a t-branch device (if anatomy suitable) Urgent patients who do not have anatomy suitable to a t-branch device or patients who are not deemed safe to wait for the device to be obtained, will undergo repair with a physician modified device.

The device is inserted into the body through two small punctures or incisions in the groin. Small stents will be inserted through the stent graft fenestrations into the major blood vessels affected by the aneurysm so that blood flow is maintained to these organs.

ELIGIBILITY:
Inclusion Criteria:

* A patient may be suitable for inclusion in the study if the patient has at least one of the following:

  1. Aortic or aortoiliac aneurysm with diameter ≥5.5 cm
  2. Aortic or aortoiliac aneurysm with a history of growth ≥1.0 cm per year, or clinical indication for aneurysm repair based on symptoms

     General Inclusion Criteria

  <!-- -->

  1. Cannot be treated with a currently available non-modified approved device
  2. Symptomatic on presentation and unsafe to wait for the time necessary to obtain a currently available non-modified approved device
  3. At least 18 years of age
  4. Not pregnant or breastfeeding
  5. Willing and able to comply with five years of follow-up
  6. Willing and able to provide informed consent prior to enrollment
  7. No systemic or local infection that may increase the risk of endovascular graft infection
  8. High risk for open surgical repair based on any of the factors below:

     a. Anatomic i. Previous abdominal surgery ii. Previous left-sided thoracotomy (if the proposed open repair would require dissection of the thoracic aorta) iii. Previous aortic surgery b. Physiologic i. ASA Category III or higher ii. Age >70 years iii. Previous myocardial infarction, coronary artery disease, or coronary artery stent iv. Coronary stress test with a reversible perfusion defect v. Congestive heart failure vi. COPD

     Exclusion Criteria:
* Exclusion Criteria Medical Exclusion Criteria

  1. Cultural objection to receipt of blood or blood products
  2. Allergy or sensitivity to stainless steel, polyester, polypropylene, solder (tin, silver), gold, or nitinol
  3. Anaphylactic reaction to contrast that cannot be adequately pre-medicated
  4. Uncorrectable coagulopathy
  5. Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
  6. Patient has active malignancy with life expectancy of less than 2 years
  7. Patient has life expectancy less than two years

Anatomical Exclusion Criteria

1. Significant occlusive disease, tortuosity, or calcification that would prevent endovascular access
2. Proximal neck length ≤25 mm
3. Proximal neck, measured outer wall to outer wall on a sectional image (CT)

   1. For use of Zenith Flex: diameter >32 mm or <18 mm
   2. For use of Zenith TX2: diameter >38 mm or <24 mm (for proximal and distal neck diameter)
4. Proximal neck angulated more than 60 degrees relative to the long axis of the aneurysm
5. Proximal neck diameter change over the length of the proximal seal zone >4 mm
6. Proximal seal site with a circumferential thrombus/atheroma
7. Iliac artery diameter, measured inner wall to inner wall on a sectional image (CT) <7.0 mm at any point along access length (prior to deployment)
8. Ipsilateral iliac artery fixation site diameter, measured inner wall on a sectional image (CT) >21 mm at distal fixation site
9. Iliac artery distal fixation site <10 mm in length
10. Non-bifurcated segment of any artery to be stented < 15 mm in length
11. Artery to be stented with a maximum diameter <3 mm or >10 mm at the vessel ostium
12. Inability to maintain at least one patent hypogastric artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-03; Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of physician modified endovascular grafts will be determined by evaluating the proportion of patients that achieve Treatment Success | 12 months post procedure
  Treatment success is a combination of technical success, and freedom at 12 months from the following: Type 1 and 3 Endoleaks, Stent migration of more than 10 mm, aortic aneurysm enlargement sac enlargement of more than 5 mm, aneurysm rupture and conversion to open repair.

SECONDARY OUTCOMES:
Incidence of Major Adverse Events | Within 30 days of the initial procedure
  Major adverse events include death, myocardial infarction, stroke, respiratory failure, paralysis, bowel ischemia, and procedural blood loss of greater than 1 liter.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Schanzer, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Health Care - University Campus, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Derived] Finnesgard EJ, Simons JP, Jones DW, Judelson DR, Aiello FA, Boitano LT, Sorensen CM, Nguyen TT, Schanzer A. Initial single-center experience using Fiber Optic RealShape guidance in complex endovascular aortic repair. J Vasc Surg. 2023 Apr;77(4):975-981. doi: 10.1016/j.jvs.2022.11.041. Epub 2022 Nov 13. PMID 36384183
- [Derived] Alqaim M, Cosar E, Crawford AS, Robichaud DI, Walz JM, Schanzer A, Simons JP. Lumbar drain complications in patients undergoing fenestrated or branched endovascular aortic aneurysm repair: Development of an institutional protocol for lumbar drain management. J Vasc Surg. 2020 Nov;72(5):1576-1583. doi: 10.1016/j.jvs.2020.02.013. Epub 2020 Apr 2. PMID 32249045
- [Derived] Schanzer A, Baril D, Robinson WP 3rd, Simons JP, Aiello FA, Messina LM. Developing a complex endovascular fenestrated and branched aortic program. J Vasc Surg. 2015 Mar;61(3):826-31. doi: 10.1016/j.jvs.2014.08.121. Epub 2015 Jan 13. PMID 25595400